CLINICAL TRIAL: NCT03691480
Title: Outpatient Management of Primary Spontaneous Pneumothorax: Pigtail Catheter With Unidirectional Valve vs. Exsufflation, Randomized Prospective Study
Acronym: PNEUM-AMBU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC17_8995_PNEUM-AMBU; 2019-A00085-52 (Other: N°ID-RCB)
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pneumothorax, Spontaneous
MeSH Terms: conditions — Pneumothorax | interventions — Ambulatory Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simple exsufflation (Experimental)
  Interventions: Procedure: simple exsufflation
- Fuhrman catheter and ambulatory care (Experimental)
  Interventions: Procedure: Fuhrman catheter and ambulatory care

INTERVENTIONS:
Procedure: simple exsufflation — simple exsufflation
  Arms: simple exsufflation
Procedure: Fuhrman catheter and ambulatory care — Fuhrman catheter and ambulatory care
  Arms: Fuhrman catheter and ambulatory care

SUMMARY:
The management of spontaneous large pneumothorax is not consensual. The current management involves the establishment of a Fuhrman catheter and an outpatient monitoring in pneumology consultation. Another alternative is widespread: simple exsufflation. However, no study has looked at the direct prospective comparison of these 2 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Episode of primary spontaneous pneumothorax wide according to the criteria

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Successful patient rates of ambulatory care | Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Jouneau, Principal Investigator — CHU Rennes
Locations (5):
- France (5):
  - CH Lorient, Lorient
  - CHU Rennes, Rennes
  - CH Sélestat, Sélestat
  - CH Saint-Malo, St-Malo
  - CHU Toulouse, Toulouse